CLINICAL TRIAL: NCT00216320
Title: A Three-Arm, Randomized Crossover Study Comparing the Innovative Neurotronics WalkAide™ System to Ankle-Foot Orthosis [AFO]
Brief Title: Efficacy of the WalkAide and AFOs for CVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovative Neurotronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WalkAide Trials
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Stroke
Keywords: electrical stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- WalkAide (Experimental): Subjects wear WalkAide for 6 weeks then cross over to AFO wear for 6 weeks
  Interventions: Device: WalkAide; Device: AFO
- Ankle Foot Orthosis (Active Comparator): Subjects wear AFO for 6 weeks then cross over to WalkAide wear for 6 weeks
  Interventions: Device: WalkAide; Device: AFO
- No Crossover (Other): Subjects wear AFO for entire 12 weeks with no crossover
  Interventions: Device: AFO

INTERVENTIONS:
Device: WalkAide — Arm 1 - Subjects wear WalkAide for 6 weeks then cross over to AFO wear for 6 weeks
  Arms: Ankle Foot Orthosis; WalkAide
Device: AFO — Arm 2 - Subjects wear AFO for 6 weeks then cross over to WalkAide wear for 6 weeks
  Arms: Ankle Foot Orthosis; WalkAide
Device: AFO — Arm 3 - Subjects wear AFO for entire 12 weeks with no crossover
  Arms: No Crossover

SUMMARY:
To assess the effectiveness of a new stimulator (WalkAide) for the treatment of foot drop. The comparison will involve physical measurements (e.g. walking speed, physiological cost index, Modified Rivermead Mobility Index, etc.) and questionnaires on the quality of life and acceptance of the technology by stroke survivors.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death in the United States and other developed countries and a major source of disability, often leading to hospitalization. Prognosis for regaining the ability to walk is good, with 64% of those initially dependent in walking regaining independence by three months. However, many gait abnormalities persist.

Reduced hip, knee and ankle excursions during swing are among the persistent gait abnormalities contributing to poor or inefficient limb clearance. This is generally referred to as "foot drop", since the foot drops or drags along the ground during the swing phase. Swing phase abnormalities can result in decreased velocity, limited endurance and an increased risk for falls. These factors can limit mobility and independence in the community. Therefore, intervention is warranted.

The conventional approach to address the poor swing limb function, specifically, insufficient ankle dorsiflexion, is the prescription of an ankle-foot orthosis (AFO). An AFO commonly limits ankle plantarflexion to enhance limb clearance during swing. An alternative approach is to stimulate the ankle dorsiflexors electrically during swing phase to reproduce motion, which can no longer be performed volitionally.

The WalkAide is a new foot drop stimulator. This small, self-contained device attaches to the leg below the knee. The WalkAide contains a number of patented features, including a tilt sensor that measures the orientation of the leg with respect to the vertical. When the leg is tilted back at the end of stance, stimulation of the common peroneal nerve is initiated. This produces flexion of the ankle and other joints (if a flexion reflex is elicited) so that the leg can clear the ground during swing. When the leg is tilted forward at the end of swing phase, the stimulus is terminated. The electrodes attach to the inside of a cuff that is molded to the leg for reproducible positioning from day to day. The device is also designed so that all operations can be done with a single hand, since hemiparesis may prevent the subject from using the other hand. Because of its enhanced features, the WalkAide is anticipated to increase walking speed and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Diagnosed with cerebrovascular accident (CVA) within the last 365 days
3. Inadequate dorsiflexion during the swing phase of gait, resulting in inadequate limb clearance
4. Medically stable for six months prior to the most recent episode of stroke resulting in hemiplegia or hemiparesis with foot drop
5. Medical clearance by the attending physician to participate in the study
6. Expectation that current medication can be maintained without drastic change for at least six months
7. Adequate stability at the ankle during stance (with stimulation)
8. Adequate cognitive and communication function to give informed consent, understand the training instructions, use the device and give adequate feedback
9. Ability to ambulate with or without an assistive device (or assistance) at least 10 meters

Exclusion Criteria:

1. Lower motor neuron injury with inadequate response to stimulation
2. History of falls greater than once a week prior to the CVA
3. Severe cardiac disease such as myocardial infarction, congestive heart failure or a demand pacemaker (or other electrical stimulator)
4. Fixed ankle contractures of five degrees of plantarflexion with knee extended
5. Moderate to normal ambulation velocity (greater than 1.2 m/s)
6. Unable to operate the device safely by self and caregiver assistance not available
7. Need for an AFO for stance control of the foot, ankle and/or knee
8. Comorbid conditions unlikely to survive one year
9. Pre-existing history of seizure disorder prior to most recent episode of CVA
10. Pre-existing pathology resulting in a significant disruption in alignment or function of the lower extremity
11. Morbid obesity that limits the subject's response to stimulation due to adipose tissue [BMI > 40]
12. Excessive dysesthetic pain secondary to neurological involvement
13. Severe hypertonicity resulting in the need for more involved orthotic strategies or pharmacological interventions (e.g. Botox)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Munin, MD, Principal Investigator — University of Pittsburgh, Department of PM&R; Sunil Hegde, MD, Principal Investigator — Huntington Rehabilitation Medicine Associates; Gerard Francisco, MD, Principal Investigator — Texas Institute of Rehabilitation Research; Richard Herman, MD, Principal Investigator — Good Samaritan Rehabilitation Institute; Thy Huskey, MD, Principal Investigator — Washington University in St. Louis, Department of Neurology; Gary Abrams, MD, Principal Investigator — University of California; San Francisco VA Medical Center
Locations (5):
- United States (5):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - San Francisco VA Medical Center, San Francisco, California
  - Washington University, St Louis, Missouri
  - University of Pittsburgh, Department of PM&R, Pittsburgh, Pennsylvania
  - Texas Institute of Rehabilitation Research, Houston, Texas

REFERENCES:
- [Result] Everaert DG, Stein RB, Abrams GM, Dromerick AW, Francisco GE, Hafner BJ, Huskey TN, Munin MC, Nolan KJ, Kufta CV. Effect of a foot-drop stimulator and ankle-foot orthosis on walking performance after stroke: a multicenter randomized controlled trial. Neurorehabil Neural Repair. 2013 Sep;27(7):579-91. doi: 10.1177/1545968313481278. Epub 2013 Apr 4. PMID 23558080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between May 2005 and December 2008 at 9 Rehabilitation centers in the USA.
Groups:
- Arm 1: WalkAide: Subjects started with the WalkAide and crossed over to the AFO after six weeks.
- Arm 2: Ankle Foot Orthosis: Subjects started with the AFO and crossed over to the WalkAide after six weeks.
- Arm 3: No Crossover: Subjects completed the entire 12 weeks period with the AFO, no crossover occurred.
Period: Phase 1 (Weeks 0 - 6)
Arm/Group | Arm 1: WalkAide | Arm 2: Ankle Foot Orthosis | Arm 3: No Crossover
Started | 43 | 39 | 30
Completed | 43 | 35 | 25
Not Completed | 0 | 4 | 5
Period: Phase 2 (Weeks 6 -12)
Arm/Group | Arm 1: WalkAide | Arm 2: Ankle Foot Orthosis | Arm 3: No Crossover
Started | 43 | 35 | 25
Completed | 38 | 31 | 24
Not Completed | 5 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: WalkAide | Arm 2: Ankle Foot Orthosis | Arm 3: No Crossover | Total
Number analyzed (Participants) | 43 | 39 | 30 | 112
Age Continuous [Mean (Standard Deviation); unit: years] | 57.1 (12.9) | 55.6 (11.9) | 58.8 (9.8) | 57.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 12 | 35
  Male | 36 | 23 | 18 | 77
Chronicity [Mean (Standard Deviation); unit: years] — Chronicity refers to the number of years since onset of stroke
  years | 6.4 (3.8) | 6.9 (3.2) | 5.8 (3.7) | 6.4 (3.6)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Subjects Who Preferred Use of WalkAide Over the Use of AFO
Description: Subjects in Arm 1 or 2 (who used both devices) were given the option to continue using WalkAide or AFO for additional 12 weeks, their preference was recorded along with reasons for preference
Time Frame: 12 weeks
Population: per protocol (completers) analysis
Measure: Number; unit: participants
Groups:
- Subjects Who Used Both WA and AFO: Subjects in arm 1 (wore WalkAide for 6 weeks followed by AFO for 6 weeks) and arm 2 (wore AFO for 6 weeks followed by WalkAide for 6 weeks)were given the option of continuing for 12 more weeks with their choice of device
Arm/Group | Subjects Who Used Both WA and AFO
Number analyzed (Participants) | 64
participants | 45
Statistical Analysis 1: Comparison: Subjects Who Used Both WA and AFO; Test type: Superiority or Other; p < .001, Chi-squared

2. Primary Outcome: Figure 8 Walking Speed Before and After Intervention.
Description: Subjects walked a 10 meter Figure 8 pattern for four minutes at fastest safe speed. This was measured under two conditions: On condition - the WA turned on or the AFO worn by the subject; off condition - The WA turned off or the AFO not worn by the subject. The endpoints were analyzed at 6, and 12 weeks
Time Frame: baseline, 6, 6.2 and 12 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1: WalkAide | Arm 2: Ankle Foot Orthosis | Arm 3: No Crossover
Number analyzed (Participants) | 38 | 31 | 24
meters/second
  Week 0 off condition | .337 (.164) | .312 (.151) | .261 (.182)
  Week 6 off condition | .432 (.207) | .377 (.166) | .303 (.195)
  Week 0 on condition | .358 (.157) | .368 (.186) | .331 (.203)
  Week 6 on condition | .456 (.205) | .428 (.179) | .366 (.205)
  Week 6.2 off condition | .446 (.216) | .383 (.162) | .303 (.195)
  Week 12 off condition | .467 (.233) | .420 (.171) | .328 (.212)
  Week 6.2 on condition | .471 (.219) | .400 (.153) | .366 (.205)
  Week 12 on condition | .520 (.236) | .436 (.172) | .388 (.208)

3. Primary Outcome: Physiological Cost Index Before and After Intervention.
Description: PCI is the difference between resting heart rate and active heart rate during walking, divided by average walking speed. This was measured under two conditions: On condition - the WA turned on or the AFO worn by the subject; off condition - The WA turned off or the AFO not worn by the subject. The endpoints were analyzed at 6, and 12 weeks
Time Frame: baseline, 6, 6.2 and 12 weeks
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Arm 1: WalkAide | Arm 2: Ankle Foot Orthosis | Arm 3: No Crossover
Number analyzed (Participants) | 33 | 27 | 17
beats/minute
  Week 0 off condition | .957 (0618) | 1.128 (.616) | 1.486 (.753)
  Week 6 off condition | .824 (.446) | .978 (.698) | 1.311 (.720)
  Week 0 on condition | .985 (.580) | .903 (.440) | 1.163 (.621)
  Week 6 on condition | .791 (.411) | .853 (.471) | 1.022 (.455)
  Week 6.2 off condition | .796 (.484) | .908 (.499) | 1.311 (.720)
  Week 12 off condition | .712 (.494) | .983 (.662) | 1.160 (.823)
  Week 6.2 on condition | .726 (.435) | .847 (.400) | 1.022 (.455)
  Week 12 on condition | .656 (.325) | .972 (.694) | .892 (.481)

4. Primary Outcome: 10 Meter Walking Speed Before and After Intervention.
Description: Subjects walked 10 meters at their fastest safe speed. This was measured under two conditions: On condition - the WA turned on or the AFO worn by the subject; off condition - The WA turned off or the AFO not worn by the subject. The endpoints were analyzed at 6, and 12 weeks
Time Frame: baseline, 6, 6.2 and 12 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arm 1: WalkAide | Arm 2: Ankle Foot Orthosis | Arm 3: No Crossover
Number analyzed (Participants) | 38 | 31 | 24
meters/second
  Week 0 off condition | .457 (.245) | .415 (.220) | .361 (.264)
  Week 6 off condition | .575 (.291) | .489 (.233) | .428 (.286)
  Week 0 on condition | .524 (.253) | .472 (.246) | .438 (.286)
  Week 6 on condition | .625 (.309) | .568 (.261) | .500 (.308)
  Week 6.2 off condition | .591 (.304) | .486 (.229) | .428 (.286)
  Week 12 off condition | .641 (.349) | .564 (.264) | .477 (.296)
  Week 6.2 on condition | .645 (.313) | .508 (.223) | .500 (.308)
  Week 12 on condition | .730 (.369) | .596 (.278) | .546 (.326)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Arm 1: All subjects used WalkAide for the first 6 weeks and AFO for the second six weeks.
- Arm 2: All subjects used AFO for the first 6 weeks and WalkAide for the second six weeks.
- Arm 3: All subjects used AFO for all 12 weeks of study.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/39 | 1/30
Other Adverse Events (participants affected / at risk) | 7/43 | 5/39 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=43) | Arm 2 (N=39) | Arm 3 (N=30)
Heart surgery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Had emergency heart surgery 9/15/06
Death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — began experiencing symptoms, went to ER and was admitted for an acute MI. Patient was discharged from the hospital and scheduled for heart surgery to remove blockage. However he then passed away suddenly, before the surgery was done
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Pt fell and fractured wrist. Subject was in teh AFO phase of Arm @ but was not wearing a study device at the time
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=43) | Arm 2 (N=39) | Arm 3 (N=30)
Skin Irritation electrodes (Skin and subcutaneous tissue disorders) | 4 (7) | 3 (4) | 0 (0) — Irritation from electrodes used with WalkAide
Skin irritation AFO (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) — tripped and fell
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — sprained ankle getting out of bed
Sinus condition (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — subject missed visit due to sinus infection
Lost consciousness (General disorders) | 1 (1) | 0 (0) | 0 (0) — Pt lost consciousness in Physical Therapy, no reason was reported
weakness and fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) — Subject was weak and fatigued, required bedrest
LE swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Subject complained of swelling not previously noted
Shoulder surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Subject had surgery for rotator cuff tear

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No